CLINICAL TRIAL: NCT00773890
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Activity of TRF-1101 on Microvascular Blood Flow, Vascular Endothelial Injury, and Vasoocclusive Pain in Patients With Sickle Cell Disease
Brief Title: TRF-1101 Assessment in Sickle Cell Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was stopped due to perceived futility because the baseline pain score in first 40 patients was too low to be able demonstrate an improvement
Sponsor: TRF Pharma, Inc (Industry)
Responsible Party: Edward Monaghan, Vice President, Clinical Operations, TRF Pharma, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1101-201
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Last update posted 2009-05-11 (Estimated); Status verified 2009-05

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRF-1101 (Experimental): Daily treatment with TRF-1101
  Interventions: Drug: TRF-1101
- Placebo (Placebo Comparator): Daily treatment with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRF-1101 — once daily treatment with 300 mg orally for 12 weeks
  Arms: TRF-1101
Drug: Placebo — Daily treatment with TRF-1101 vehicle for 12 weeks
  Arms: Placebo

SUMMARY:
This study is designed to assess the safety, tolerability, and activity of TRF-1101 on microvascular blood flow, vascular endothelial injury, and vasoocclusive pain associated with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older at the time of informed consent;
* Have a diagnosis of homozygous sickle cell anemia or sickle cell-beta° thalassemia;
* Have had 2 - 10 documented pain crises in the past year (pain crises are defined as visits to a medical clinic, Emergency Department or hospital, being bedridden and requiring constant analgesia at home for at least three days, or having a three-day interruption of life's activities [i.e., school, work, planned leisure activity] because of pain);
* If female and of child bearing potential, have a negative serum or urine pregnancy test and be using an effective birth-control method with a history of reliability for the individual patient (use of mifepristone is not allowed);
* Be properly informed of the nature and risks of the clinical investigation, be willing and able to comply with all clinical investigation-related procedures and assessments, and sign an Institutional Review Board (IRB) approved Informed Consent Form prior to entering the clinical investigation.

Exclusion Criteria:

* Have a history of abnormal bleeding, stroke, moya moya vascular malformations, or any other contraindication to anticoagulation;
* Be currently taking anticoagulant or thrombolytic medication;
* Be currently taking an endothelin receptor antagonist, e.g., bosentan (Tracleer®);
* Have a known sensitivity or allergy to heparin or related drugs;
* Have a history of thrombocytopenia (platelet count < 100 x 103/mm3) induced by heparin or related drugs;
* Have had fewer than 2 documented pain crises in the past year;
* Have had a pain crisis within one month of screening or randomization;
* If currently on or recently discontinued hydroxyurea treatment, have initiated or discontinued treatment or changed regimen within the past 6 months;
* Have had a transfusion within last 120 days or have HbA% > 15% from prior transfusion;
* Creatinine levels > 1.53 mg/dL (135 umol/L);
* ALT levels ≥ 3 times normal;
* Platelet count < 100 x 103/mm3;
* INR > 2.0;
* Be unable to tolerate oral medications;
* Have unreliable venous access;
* Be noncompliant with regular care;
* Have a positive pregnancy test, be currently lactating, or be trying to become pregnant;
* Have participation in an investigational drug or medical device study within previous 30 days;
* Have any other condition or circumstance that in the opinion of the Investigator makes the patient a poor candidate for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
endothelial cell injury/inflammation | Throughout trial

SECONDARY OUTCOMES:
Microvascular blood flow and trends in frequency of vasoocclusive pain | throughout trial

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Embury, M.D., Study Director — TRF Pharma, Inc
Locations (6):
- United States (6):
  - Howard University, Washington D.C., District of Columbia
  - Medical College of Georgia, Augusta, Georgia
  - University of Illinios Medical Center, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - Wayne State University Medical Center, Detroit, Michigan
  - University of North Carolina, Chapel Hill, North Carolina